CLINICAL TRIAL: NCT02161822
Title: A Single Arm, Phase II Study of Neoadjuvant Chemoradiotherapy With Capecitabine Plus Simvastatin in Locally Advanced Rectal Cancer Patients
Brief Title: Capecitabine Plus Simvastatin in Locally Advanced Rectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-03-056
Record Dates: First submitted 2014-05-30; First posted 2014-06-12 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Adenocarcinoma of Rectum
Keywords: locally advanced rectal cancer, neoadjuvant chemoradiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Simvastatin (Experimental): single arm : Simvastatin
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — simvastatin 80mg qd for 5weeks
  Other Names: Zocor tab

SUMMARY:
Statins are widely used as lipid-lowering agents to lower cardiovascular risk with a favorable safety profile. In our recent in vitro study, the addition of simvastatin to chemoradiotherapy with 5-FU showed synergistic anticancer effect in various colon cancer cells (unpublished data). So we planned this study to investigate the synergistic effect of simvastatin combined with capecitabine and radiotherapy in locally advanced rectal cancer patients.

DETAILED DESCRIPTION:
1. Primary Objective: pathologic complete response rate
2. Secondary Objectives:

   1. rate of sphincter-sparing surgical procedure
   2. rate of R0 resection
   3. disease-free survival
   4. overall survival
   5. pattern of failure
   6. safety and toxicity
   7. lipid lowering effect of simvastatin

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed adenocarcinoma of rectum
* AJCC/UICC clinical stages of cT3-4 or cN+
* age ≥ 20 years
* ECOG performance status 0-1
* No prior chemotherapy and radiotherapy
* Adequate major organ functions as following:
* Written informed consent
* Willing and able to comply the protocol

Exclusion Criteria:

* Prior statins therapy within 1-year from the date of study entry
* Uncontrolled or severe cardiovascular disease :

New York Heart Association class III or IV heart disease Unstable angina or myocardial infarction within the past 6 months History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality.

* Past or current history (within the last 5 years prior to treatment start) of other malignancies except rectal cancer (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible)
* Uncontrolled systemic illness such as DM, hypertension, hypothyroidism and infection
* Pregnant nursing women (women of reproductive potential have to agree to use an effective contraceptive method)
* Patients with CPK > 5 X ULN at baseline
* Concomitant use with clarithromycin, erythromycin, itraconazole, ketoconazole, nefazodone, telithromycin, gemfibrozil, cyclosporine, danazol, amiodarone, verapamil

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | average of 5 weeks
  pathologic complete response ratewill be shown with 95% confidence intervals

SECONDARY OUTCOMES:
rate of sphincter-sparing surgical procedure | average of 5 weeks
  rate of sphincter-sparing surgical procedure
rate of R0 resection | average of 5 weeks
  rate of R0 resection (N-60)
disease-free survival | assessed up to 60 months
  disease-free survival
overall survival | assessed up to 60 months
  Time from randomization to death or last follow-up
pattern of failure | assessed up to 60 months
  Sphincter preservation
safety and toxicity | assessed up to 6 months
  Response rate according to RECIST 1,1 guideline will also be evaluated
lipid lowering effect of simvastatin | assessed up to 6 months
  Total cholesterol, LDL-cholesterol records. (2weeks)

CONTACTS AND LOCATIONS:
Overall Officials: woon ki kang, professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided